CLINICAL TRIAL: NCT01298180
Title: Is There a Sensibility Increased in the Growth Hormone at Child With Prader-Willi Syndrome?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0811601; National PHRC 2008 (Other Grant/Funding Number: PHRC 2008)
Record Dates: First submitted 2009-11-06; First posted 2011-02-17 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Prader-Willi Syndrome; Growth Hormone Deficiency
Keywords: Prader-Willi Syndrome; Growth Hormone Deficiency
MeSH Terms: conditions — Prader-Willi Syndrome; Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone; Absorptiometry, Photon; Hematologic Tests; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- SPW (Experimental): Children presenting a Prader-Willi Syndrome
  Interventions: Drug: Growth hormone (Genotonorm® or Omnitrope®); Procedure: DEXA, blood tests, H.G.P.O, osseous age.
- GHD (Experimental): Patient deficient in Growth Hormone
  Interventions: Drug: Growth hormone (Genotonorm® or Omnitrope®); Procedure: DEXA, blood tests, H.G.P.O, osseous age.
- SPW-B (Experimental): Patient with Prader-Willi Syndrome who has Biopsy
  Interventions: Drug: Growth hormone (Genotonorm® or Omnitrope®); Procedure: DEXA, blood tests, H.G.P.O, osseous age.; Procedure: biopsy
- T (Experimental): Patient Control
  Interventions: Procedure: biopsy
- SPW-GH-B (Experimental): Patient with Prader-Willi Syndrome taking growth Hormone and who has biopsy
  Interventions: Procedure: biopsy

INTERVENTIONS:
Drug: Growth hormone (Genotonorm® or Omnitrope®) — drug : the treatment will be begun in progressive dose by beginning by ¼ of the dose the first week, then ½ of the dose the second week, then 3/4 of the dose the third week and total dose the fourth week.
  Arms: GHD; SPW; SPW-B
Procedure: DEXA, blood tests, H.G.P.O, osseous age. — SPW, GHD, SPW-B :
  blood tests : centralized dosage H.G.P.O : adjusted to children's age.
  Arms: GHD; SPW; SPW-B
Procedure: biopsy — Biopsy : Cutaneous and fat tissue biopsy.
  Arms: SPW-B; SPW-GH-B; T

SUMMARY:
The purpose of this study is to estimate the sensibility at the growth hormone in vivo at the children presenting a Prader-Willi syndrome (SPW) in comparison with children presenting a deficit in growth hormone (GHD).

DETAILED DESCRIPTION:
Estimate the sensibility at the growth hormone in vivo at the children presenting a Prader-Willi syndrome (SPW) in comparison with children presenting a deficit in growth hormone (GHD) by the measure of the circulating rates of IGF-I under treatment.

ELIGIBILITY:
Inclusion Criteria:

1. SPW and SPW-B :

   * Female or male child of age > or = 1 year
   * Child naïve of treatment by GH and that must begin a treatment with GH
   * Child covered by a national insurance scheme or an equivalent
   * Signature of the informed consent by one of both holders of the parental authority
2. GHD :

   * Female or male child of age > or = 1 year
   * Child paired for the age (+/-on 1 year) and for the sex with regard to the group SWP
   * Child presenting a GH* deficiency defined by :

   Growth criteria of size (size) < 2 DS) Criteria of speed of growth (speed of growth < 1 DS over the last year) 2 tests of pharmacological stimulation of GH with peak GH max < 20 mUI
   * Child naïve of treatment by GH and that must begin a treatment with GH
   * Child covered by a national insurance scheme or an equivalent
   * Signature of the informed consent by one of both holders of the parental authority * The deficit in GH can be isolated or associated with one or several other hormonal deficits: deficit in TSH, deficit in ACTH, deficit in LH-FSH, deficit in prolactin. The child GHD can thus receive other treatments associated with the growth hormone.
3. T : controls

   * Female or male child of age > or = 1 year
   * Child paired for the age (+/-on 1 year) and for the sex with regard to the group SWP
   * Child hospitalized at the hospital of the children of the University Hospital of Toulouse for a programmed surgical operation
   * Child covered by a national insurance scheme or an equivalent
   * Signature of the informed consent by one of both holders of the parental authority
4. SPW-GH-B :

   * Female or male child of age > or = 1 year
   * Child hospitalized for a programmed surgical operation
   * Child covered by a national insurance scheme or an equivalent
   * Child treated with GH for at least 3 month
   * Signature of the informed consent by one of both holders of the parental authority

Exclusion Criteria:

1. SPW and GHD

   * Child presenting a contraindication to the taking of growth hormone :
   * Growth cartilage welded
   * Tumoral pathology in process of evolution
   * Corticosteroid therapy (not substitute)
   * Allergy known about solvent
   * Badly balanced diabetes
   * Child presenting a hypersensitivity to the active principle or to one of the excipients of Genotonorm ® or Omnitrope ®
   * Child presenting a severe obesity (defined by a report weight / size > 200 %)
   * Child presenting clinical signs ENT (snores associated with a hypertrophy of the adenoids vegetations and\or the tonsils)
   * Child presenting clinical signs evoking a respiratory illness of the sleep (night-respiratory snores, respiratory breaks during the sleep)
2. SPW-B:

   * Child presenting a hypersensitivity to the local anaesthetic with amide connecion
   * Child presenting a hypersensitivity to the components of the bandage Emlapatch®
   * Child presenting a hypersensitivity to one of the components of the lidocaïne aguettant without conservative®
   * Child presenting a porphyria
   * Child presenting a congenital methemoglobinemia
   * Child presenting a contraindication to Meopa : patients requiring a ventilation in pure oxygen, intracranial High blood pressure, Any change of the state of consciousness, preventing the cooperation of the patient, Pneumothorax, Bubbles of emphysema, Gaseous embolism, Accident of dive, abdominal gaseous Distension, Patient having received recently an ophthalmic gas (SF6, C3F8, C2F6) used in the eye surgery as long as persists a bubble of gas inside the eye and at least during a period of 3 months. Grave postoperative complications can arise in touch with the increase of the pressure intraocular, facial Traumatism interesting the region of application of the mask
3. T : controls

   * Chronicle pathology in which an abnormality of growth would be involved
   * Other hormonal abnormalities
   * Children receiving a treatment on the long range, corticosteroid therapy in particular, being able to interfere with the sensibility to GH or to the insulin
   * Holder of the parental authority under supervision, guardianship or under protection of justice
   * Participation in another study simultaneously at this one

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measure of the circulating rates of IGF-I under treatment. | Before starting treatment: baseline (J0)
Measure of the circulating rates of IGF-I under treatment. | 1 month (M1)
Measure of the circulating rates of IGF-I under treatment. | 3 month (M3)
Measure of the circulating rates of IGF-I under treatment. | 6 month (M6)
Measure of the circulating rates of IGF-I under treatment. | 1 year (M12)

SECONDARY OUTCOMES:
Measure of the circulating rate of IGFBP-3, GHBP, ghrelin and apelin. | Before starting treatment (J0)
Measure of physical composition's variation. | Before starting treatment (J0)
Measure of blood sugar level, H.G.P.O., and hyperglycaemia. | Before starting treatment (J0)
Measure of the sensibility at the growth hormone in vitro, on fibroblasts and adipocytes obtained by biopsy. | Before starting treatment (J0)
Measure of the circulating rate of IGFBP-3, GHBP, ghrelin and apelin. | 3 months (M3)
Measure of the circulating rate of IGFBP-3, GHBP, ghrelin and apelin. | 6 months (M6)
Measure of the circulating rate of IGFBP-3, GHBP, ghrelin and apelin. | 1 year (M12)
Measure of physical composition's variation. | 3 months (M3)
Measure of physical composition's variation. | 6 months (M6)
Measure of physical composition's variation. | 1 year (M12)
Measure of blood sugar level, H.G.P.O., and hyperglycaemia. | 3 months (M3)
Measure of blood sugar level, H.G.P.O., and hyperglycaemia. | 6 months (M6)
Measure of blood sugar level, H.G.P.O., and hyperglycaemia. | 1 year (M12)
Measure of the sensibility at the growth hormone in vitro, on fibroblasts and adipocytes obtained by biopsy. | 3 months (M3)
Measure of the sensibility at the growth hormone in vitro, on fibroblasts and adipocytes obtained by biopsy. | 6 months (M6)
Measure of the sensibility at the growth hormone in vitro, on fibroblasts and adipocytes obtained by biopsy. | 1 year (M12)

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (26):
- France (26):
  - CHU Amiens Hôpital Nord Service Pédiatrie - Place Victor Pauchet, Amiens
  - CHU Angers - 4 rue Larrey, Angers
  - CHG Avignon - 305, rue Raoul Follereau, Avignon
  - CHU Besançon Hôpital Saint Jacques - 2 Place Saint Jacques, Besançon
  - CHU Bordeaux Hôpital Pellegrin Service endocrinologie de l'enfant - Place Amélie Raba Léon, Bordeaux
  - CHU Brest Département de Pédiatrie - 5, ave Foch, Brest
  - CHU Dijon Service de pédiatrie - 2, Bd Maréchal de lattre de Tassigny, Dijon
  - CHU Grenoble Service de pédiatrie - BP 217, Grenoble
  - CHU La Rochelle Service de Pédiatrie - Rue du Dr Schweitzer, La Rochelle
  - CHRU Lille Hôpital Jeanne de Flandre service de Pédiatrie, Lille
  - CHU Limoges Hôpital Mère Enfant Service Pédiatrie - 8, ave du Larrey, Limoges
  - CHU Lorient Hôpital du Scorff Pôle Femme Mère Enfant - Rue Guiguen, Lorient
  - CHU Lyon Hôpital Debrousse service Pédiatrie, Lyon
  - AP-HM Hôptal La Timone Service de Pédiatrie Mutidisciplinaire, Marseille
  - CHU Montpellier Hôpital Arnaud de Villeneuve - 371 ave du doyen Gaston Giraud, Montpellier
  - CHU Nantes Hôpital Mère Enfant Service de Pédiatrie, Nantes
  - CHU Nice Hôpital Archet 2 - 151 route Saint Antoine de Ginestière, Nice
  - AP-HP Hôpital Necker Enfants Malades Service d'endocrinologie pédiatrique - 149 route de Sèvres, Paris
  - CHU Poitiers Service de Pédiatrie - Rue de la Miléterie, Poitiers
  - CHU Reims Service de Pédiatrie - 47, rue Cognacq-Jay, Reims
  - CHU Rouen Hôpital Nicolle - 1, rue de Germont, Rouen
  - CHU Saint-Etienne Hôpital Nord Service de Pédiatrie, Saint-Etienne
  - CHU Strasbourg Hôpital Haute-Pierre - Avenue Molière, Strasbourg
  - CHU Toulouse Hôpital des Enfants Service d'endocrinologie - 330 ave de Grande Bretagne, Toulouse
  - CHRU Tours Centre de Pédiatrie Gatien de Clocheville, Tours
  - Hôpital d'Enfants - Rue Morvan, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Cadoudal T, Buleon M, Sengenes C, Diene G, Desneulin F, Molinas C, Eddiry S, Conte-Auriol F, Daviaud D, Martin PG, Bouloumie A, Salles JP, Tauber M, Valet P. Impairment of adipose tissue in Prader-Willi syndrome rescued by growth hormone treatment. Int J Obes (Lond). 2014 Sep;38(9):1234-40. doi: 10.1038/ijo.2014.3. Epub 2014 Jan 10. PMID 24406482
- [Result] Eddiry S, Diene G, Molinas C, Salles J, Auriol FC, Gennero I, Bieth E, Skryabin BV, Rozhdestvensky TS, Burnett LC, Leibel RL, Tauber M, Salles JP. SNORD116 and growth hormone therapy impact IGFBP7 in Prader-Willi syndrome. Genet Med. 2021 Sep;23(9):1664-1672. doi: 10.1038/s41436-021-01185-y. Epub 2021 May 26. PMID 34040195
- [Result] Bieth E, Eddiry S, Gaston V, Lorenzini F, Buffet A, Conte Auriol F, Molinas C, Cailley D, Rooryck C, Arveiler B, Cavaille J, Salles JP, Tauber M. Highly restricted deletion of the SNORD116 region is implicated in Prader-Willi Syndrome. Eur J Hum Genet. 2015 Feb;23(2):252-5. doi: 10.1038/ejhg.2014.103. Epub 2014 Jun 11. PMID 24916642